CLINICAL TRIAL: NCT05891171
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of AB598 Monotherapy and Combination Therapy in Participants With Advanced Malignancies
Brief Title: Study of AB598 Monotherapy and Combination Therapy in Participants With Advanced Cancers
Acronym: ARC-25
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-25
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Cancer; Advanced Malignancies; Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Gastroesophageal-junction Cancer (GEJ); Head and Neck Squamous Cell Carcinoma (HNSCC); Non-Small Cell Lung Cancer (NSCLC); Ovarian Cancer; Renal Cell Carcinoma (RCC); Triple Negative Breast Cancer (TNBC)
Keywords: AB598; AB122; Zimberelimab
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms | interventions — zimberelimab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Cohort 1 (Experimental): Participants will receive AB598 intravenous (IV) infusion once every 3 weeks
  Interventions: Drug: AB598
- Dose Escalation Cohort 2 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Dose Escalation Cohort 3 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Dose Escalation Cohort 4 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Pharmacodynamic Cohort 1 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Pharmacodynamic Cohort 2 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Pharmacodynamic Cohort 3 (Experimental): Participants will receive AB598 IV infusion once every 3 weeks
  Interventions: Drug: AB598
- Dose Expansion Gastric/GEJ Cancer (phase 1b) (Experimental): Participants will receive AB598 IV infusion every 2 weeks in combination with zimberelimab and FOLFOX (oxaliplatin, leucovorin, fluorouracil)
  Interventions: Drug: AB598; Drug: Zimberelimab; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: AB598 — Administered as specified in the treatment arm
Drug: Zimberelimab — Administered as specified in the treatment arm
  Other Names: AB122
  Arms: Dose Expansion Gastric/GEJ Cancer (phase 1b)
Drug: Fluorouracil — Administered as specified in the treatment arm
  Arms: Dose Expansion Gastric/GEJ Cancer (phase 1b)
Drug: Leucovorin — Administered as specified in the treatment arm
  Arms: Dose Expansion Gastric/GEJ Cancer (phase 1b)
Drug: Oxaliplatin — Administered as specified in the treatment arm
  Arms: Dose Expansion Gastric/GEJ Cancer (phase 1b)

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AB598 in participants with advanced malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) guidance
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Prior systemic radiation or whole brain radiation therapy must have been completed at least 4 weeks before investigational product (IP) administration. Other palliative radiotherapy must be completed 2 weeks before investigational product administration, if radiation therapy-related AEs have resolved to Grade ≤ 1.
* Monotherapy-specific criteria for dose escalation and PD cohorts:

  * Dose Escalation: Participants may have any pathologically confirmed advanced or metastatic solid tumor for which standard therapy has proven ineffective, intolerable, or is considered inappropriate.
  * Pharmacodynamic Cohorts: Participants may have any pathologically confirmed advanced or metastatic solid tumors for which standard therapy has proven ineffective, intolerable, or is considered inappropriate. Participants must be able to undergo collection of a fresh frozen biopsy during screening, as well as provide an on-treatment fresh frozen biopsy.
* Dose Expansion cohort criteria:

  * Histologically confirmed, documented diagnosis of HER2-negative locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma.
  * No prior systemic treatment for locally advanced unresectable or metastatic disease.
  * Cannot have progressed within 6 months of prior platinum-based chemotherapy for earlier stage disease.

Key Exclusion Criteria:

* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of initiation of study
* Underlying medical conditions or AEs that, in the investigator or sponsor's opinion, will make the administration of the study drugs hazardous
* Any active or documented history of autoimmune disease including but not limited to inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis, within 3 years of the first dose of study treatment
* History of trauma or major surgery within 28 days prior to the first dose of study drug
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressant medication during study treatment with certain protocol specified exceptions

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 2 years
Dose Escalation Cohorts: Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to 2 years

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Administration ("0") to the Time That the Drug is No Longer Present in the Body ("infinity") (AUC 0-inf) in Whole Blood and Plasma | Predose, Up to 4 hours post dose
Maximum Concentration (Cmax) in Whole Blood and Plasma | Predose, Up to 4 hours post dose
Time to Maximum Concentration (Tmax) in Whole Blood and Plasma | Predose, Up to 4 hours post dose
Number of Participants Who Test Positive for Antidrug Antibodies (ADAs) to AB598 | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
Dose Expansion Cohort: Duration of Response (DOR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (15):
- United States (11):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Lake City Cancer Care, LLC., Lake City, Florida
  - Affinity Health Hope and Healing Cancer Services, LLC, Hinsdale, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Gabrail Cancer Center (GCC) Canton Facility, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Next Oncology Dallas, Irving, Texas
  - Next Oncology Virginia, Fairfax, Virginia
- Australia (2):
  - Adelaide Cancer Research, Adelaide
  - Queen Elizabeth Hospital, Adelaide
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-25 - Public website — https://trials.arcusbio.com/study/?id=ARC-25